CLINICAL TRIAL: NCT00036335
Title: Duloxetine Hydrochloride (LY248686) Protocol F1J-US-HMCB Duloxetine Once-Daily Dosing Versus Placebo in Patients With Major Depression and Pain
Brief Title: Subject Information and Consent Form F1J-US-HMCB Duloxetine Once-Daily Dosing Versus Placebo in Patients With Major Depression and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6353; F1J-US-HMCB
Record Dates: First submitted 2002-05-08; First posted 2002-05-10 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Depression; Pain
Keywords: depression; pain; blues; sadness; aches
MeSH Terms: conditions — Depression; Pain | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride

SUMMARY:
The purposes of this study are to determine whether an investigational drug can help patients suffering from major depression with pain symptoms, and gather data on the safety of the investigational drug including any side effects that might be associated with it.

ELIGIBILITY:
Inclusion Criteria:

* You must be suffering from symptoms of depression for at least the past 2 weeks (sadness, loss of interest in daily activities, feelings of hopelessness or guilt, sleeplessness or lack of energy)
* You must have pain symptoms with no known cause, such as unexplainable, head, chest, or back pain, overall aches and pains, or other unexplainable pains.
* You need to be available to visit a doctor's office about once a week for 10 weeks.

Exclusion Criteria:

* You are a woman and are pregnant or breastfeeding.
* You have a current or previous diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder.
* You have had a primary diagnosis of an anxiety disorder within the past 6 months.
* You have a history of alcohol or drug dependence or abuse within the past 6 months.
* You have a serious medical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286
Dates: Start 2002-03; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Peoria, Arizona
  - Burbank, California
  - Fresno, California
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Oakbrook Terrace, Illinois
  - Springfield, Illinois
  - Glen Burnie, Maryland
  - Farmington Hills, Michigan
  - Nashua, New Hampshire
  - Clementon, New Jersey
  - Moorestown, New Jersey
  - Albany, New York
  - Olean, New York
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Woodstock, Vermont
  - Richmond, Virginia
  - Seattle, Washington
  - Brown Deer, Wisconsin

REFERENCES:
- [Derived] Harada E, Kato M, Fujikoshi S, Wohlreich MM, Berggren L, Tokuoka H. Changes in energy during treatment of depression: an analysis of duloxetine in double-blind placebo-controlled trials. Int J Clin Pract. 2015 Oct;69(10):1139-48. doi: 10.1111/ijcp.12658. Epub 2015 May 16. PMID 25980552
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392